CLINICAL TRIAL: NCT01403051
Title: A Prospective, Randomized, Double-Blind Phase II Trial of High-Dose Vitamin D and Calcium for Bone Health in HIV-Infected Individuals Initiating Highly Active Antiretroviral Therapy (HAART)
Brief Title: High Dose Vitamin D and Calcium for Bone Health in Individuals Initiating HAART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5280; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: EFV/FTC/TDF plus vitamin D3 and calcium carbonate (Experimental): Participants were administered FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (Atripla), calcium carbonate and vitamin D3 4000 IU.
  Interventions: Drug: EFV/FTC/TDF; Drug: Calcium Carbonate; Drug: Vitamin D3
- Arm B: EFV/FTC/TDF plus vitamin D placebo and calcium placebo (Experimental): Participants were administered FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (Atripla), a placebo for calcium carbonate, and a placebo for vitamin D3.
  Interventions: Drug: EFV/FTC/TDF; Drug: Placebo for calcium carbonate; Drug: Placebo for vitamin D3

INTERVENTIONS:
Drug: EFV/FTC/TDF — FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (Atripla) 600 mg/200 mg/ 300 mg tablet taken orally once daily at bedtime on an empty stomach.
  Other Names: Atripla
Drug: Calcium Carbonate — Calcium carbonate 500 mg tablet taken orally twice daily with food for 48 weeks.
  Arms: Arm A: EFV/FTC/TDF plus vitamin D3 and calcium carbonate
Drug: Vitamin D3 — One Vitamin D3 4000 IU capsule taken orally once daily with food for 48 weeks.
  Arms: Arm A: EFV/FTC/TDF plus vitamin D3 and calcium carbonate
Drug: Placebo for calcium carbonate — A placebo for calcium carbonate twice daily taken orally as one x 0 mg tablets with food for 48 weeks
  Arms: Arm B: EFV/FTC/TDF plus vitamin D placebo and calcium placebo
Drug: Placebo for vitamin D3 — A placebo for vitamin D3 once daily taken orally as one capsule with food for 48 weeks.
  Arms: Arm B: EFV/FTC/TDF plus vitamin D placebo and calcium placebo

SUMMARY:
This study was done with people who were infected with HIV and needed to start treatment for their HIV disease. The purpose of this study is to see if taking vitamin D and calcium will help prevent the bone loss that sometimes happens when people start HIV treatment. For this study, the following HIV treatment (or HAART) were provided in the form of a single tablet that contains three different drugs: efavirenz/emtricitabine/tenofovir (EFV/FTC/TDF). These drugs are approved by the FDA to treat HIV infection. The HIV treatment provided is common for people who are taking HIV drugs for the first time. The risks seen with this HIV treatment are the same that you would encounter when taking these drugs outside of the study. The lists of risks of this HIV treatment are included in this document because the drugs are provided by the study, not because the drugs are being tested. The purpose of the study is only to look at the impact of high doses of vitamin D and calcium in preventing bone loss. There are no study objectives related to HIV treatment (EFV/FTC/TDF).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* No evidence of any exclusionary resistance mutations based on results from any genotype assay from any laboratory that has a CLIA (Clinical Laboratory Improvement Amendments) certification or its equivalent. Results must be available from testing any time in the past or must be obtained prior to entry and reviewed by the site investigator.
* ARV drug-naïve (<=10 days of ART at any time prior to entry) and no ARV drugs taken within the past 30 days.
* CD4+ cell count of any value obtained within 90 days prior to study entry at any laboratory that has a CLIA certification or its equivalent.
* HIV-1 RNA >1000 copies/mL obtained within 90 days prior to study entry at any laboratory that has a CLIA certification or its equivalent.
* Certain laboratory values obtained within 30 days prior to entry (as indicated in section 4.1.6 of the protocol.
* Serum calcium < 10.5 mg/dL within 30 days prior to entry.
* For women of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to initiating study medications.
* Subjects must refrain from participating in a conception process (i.e., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) and if participating in sexual activity that could lead to pregnancy, the subject/partner must use at least two of the reliable forms of contraceptive listed in section 4.1.9 of the protocol.
* 25-OH vitamin D >=10 ng/mL and <75 ng/mL.
* Ability and willingness of subject or legally authorized representative to provide informed consent.

Exclusion Criteria:

* Current or prior use of bisphosphonate therapy.
* Use of vitamin D supplements greater than 800 IU/day within 30 days prior to entry.
* Use of calcium supplements greater than 500 mg/day within 30 days prior to entry.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulations.
* Any oral, intravenous, or inhaled steroids within the 30 days prior to enrollment(intranasal steroid use is allowed).
* Use of androgenic hormones or growth hormones.
* Receipt of systemic cytotoxic chemotherapy within 30 days prior to entry.
* Pregnancy or currently breastfeeding.
* Documentation of acute opportunistic infections within 30 days prior to entry.
* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to entry.
* Weight >300 lbs (exceeds weight limit of DXA scanners).
* History of nephrolithiasis (kidney stones).
* History of osteoporosis (as documented by DXA scan) or fragility fracture.
* Clinically active thyroid disease (use of thyroid hormone replacement therapy permitted but TSH must be in normal range).
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric illness.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar (Turner) Overton, MD, Study Chair — Alabama Therapeutics CRS; Michael T Yin, MD, MS, Study Chair — HIV Prevention & Treatment CRS
Locations (39):
- United States (38):
  - Alabama Therapeutics CRS (5801), Birmingham, Alabama
  - Usc Crs (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Stanford CRS (501), Palo Alto, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Georgetown University CRS (GU CRS) (1008), Washington D.C., District of Columbia
  - The Ponce de Leon Ctr. CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush University Medical Center (2702), Chicago, Illinois
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS (103), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - New Jersey Medical School-Adult Clinical Research Ctr. CRS (31477), Newark, New Jersey
  - Cornell CRS (7804), New York, New York
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - HIV Prevention & Treatment CRS (30329), New York, New York
  - AIDS Care CRS (1108), Rochester, New York
  - University of Rochester ACTG CRS (1101), Rochester, New York
  - Bronx-Lebanon Hosp. Ctr. CRS (31469), The Bronx, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Duke University Medical Center Adult CRS (1601), Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - MetroHealth CRS (2503), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS (2951), Providence, Rhode Island
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Trinity Health and Wellness Center CRS (31443), Dallas, Texas
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Derived] Yin MT, Chan ES, Brown TT, Kinslow J, Martinson J, Landay A, Melbourne KM, Ribaudo HJ, Overton ET; A5280 Study Team. Vitamin D does not modulate immune-mediated bone loss during ART initiation. Antivir Ther. 2019;24(5):355-362. doi: 10.3851/IMP3316. PMID 31085814
- [Derived] Yin MT, Chan ES, Brown TT, Tebas P, McComsey GA, Melbourne KM, Napoli A, Hardin WR, Ribaudo HJ, Overton ET; A5280 Study Team. Racial differences in calculated bioavailable vitamin D with vitamin D/calcium supplementation. AIDS. 2017 Nov 13;31(17):2337-2344. doi: 10.1097/QAD.0000000000001621. PMID 28832406
- [Derived] Overton ET, Chan ES, Brown TT, Tebas P, McComsey GA, Melbourne KM, Napoli A, Hardin WR, Ribaudo HJ, Yin MT. Vitamin D and Calcium Attenuate Bone Loss With Antiretroviral Therapy Initiation: A Randomized Trial. Ann Intern Med. 2015 Jun 16;162(12):815-24. doi: 10.7326/M14-1409. PMID 26075752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A5280 opened under version 1.0 on September 15, 2011, and the first subject was randomized on September 26, 2011. Accrual to the study closed on March 2, 2012, with a total of 167 subjects enrolled from 39 sites within the US.
Pre-assignment Details: Subjects were randomized with a 1:1 ratio at enrollment.
Groups:
- Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF: The participants were administered vitamin D3, calcium carbonate and FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (Atripla).
  Vitamin D3: One Vitamin D3 4000 IU capsule taken orally once daily with food for 48 weeks.
  Calcium Carbonate: Calcium carbonate 500 mg tablet taken orally twice daily with food for 48 weeks.
  Atripla: FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF) 600 mg/200 mg/ 300 mg tablet taken orally once daily at bedtime on an empty stomach.
- Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF: The participants were administered a placebo for vitamin D3, a placebo for calcium carbonate, and FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (Atripla)
  Placebo for vitamin D3: A placebo for vitamin D3 once daily taken orally as one capsule with food for 48 weeks.
  Placebo for calcium carbonate: A placebo for calcium carbonate twice daily taken orally as one x 0 mg tablets with food for 48 weeks
  Atripla: FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF) 600 mg/200 mg/ 300 mg tablet taken orally once daily at bedtime on an empty stomach.
Period: Overall Study
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Started | 81 | 86
Initiated Study Treatment | 81 | 86
Completed | 71 | 80
Not Completed | 10 | 6
Not completed — Protocol Violation | 2 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Population: Includes only subjects who did not have eligibility violations
Groups:
- Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF: The participants were administered a placebo for vitamin D3, a placebo for calcium carbonate, and FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (Atripla).
  Placebo for vitamin D3: A placebo for vitamin D3 once daily taken orally as one capsule with food for 48 weeks.
  Placebo for calcium carbonate: A placebo for calcium carbonate twice daily taken orally as one x 0 mg tablets with food for 48 weeks
  Atripla: FDC efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF) 600 mg/200 mg/ 300 mg tablet taken orally once daily at bedtime on an empty stomach.
- Total: Total of all reporting groups
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF | Total
Number analyzed (Participants) | 79 | 86 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 85 | 161
  >=65 years | 3 | 1 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [28 to 47] | 31 [25 to 44] | 33 [26 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 72 | 77 | 149
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 28 | 33 | 61
  Black Non-Hispanic | 24 | 30 | 54
  Hispanic (Regardless of Race) | 23 | 18 | 41
  Asian, Pacific Islander | 2 | 5 | 7
  American Indian, Alaskan Native | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 79 | 86 | 165
HIV-1 RNA level [Median (Inter-Quartile Range); unit: log10 copies/mL] — Entry HIV-RNA level (log10 copies/mL)
  log10 copies/mL | 4.5 [4.1 to 5.1] | 4.5 [4.0 to 5.1] | 4.5 [4.1 to 5.1]
CD4 count [Median (Inter-Quartile Range); unit: cells/mm3] — Entry total CD4 count (cells/mm3)
  cells/mm3 | 339 [230 to 500] | 342 [232 to 454] | 341 [230 to 490]

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change From Baseline in Bone Mineral Density (BMD) at Total Hip
Description: The efficacy endpoint is the percent change from baseline to week 48 in bone mineral density (BMD) at total hip (as measured by DXA scan)
Time Frame: Weeks 0 and 48
Population: The primary analysis is intent-to-treat (ITT) which is limited to eligible subjects who have baseline and week 48 follow-up regardless of treatment change or discontinuation.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 65 | 77
percentage change | -1.46 [-3.16 to -0.40] | -3.19 [-5.12 to -1.02]
Statistical Analysis 1: Comparison: Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF vs Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF; The study was sized to have 80% power to detect a 2 % difference in BMD of the hip from baseline to week 48; Test type: Superiority or Other; p = 0.001, Stratified Wilcoxon rank sum test — 2-sided test with type I error rate of 5%, not adjusted for multiple comparisons; Stratified Wilcoxon rank sum test for differences between the two treatment groups, stratified by the screening 25-OH vitamin (<=20 vs. >20 ng/mL)

2. Secondary Outcome: The Percent Change From Baseline in Bone Mineral Density (BMD) at Spine
Description: The percent change from baseline to week 48 in bone mineral density (BMD) at spine as measured by DXA scan
Time Frame: Weeks 0 and 48
Population: This analysis is intent-to-treat (ITT) which is limited to eligible subjects who have baseline and week 48 follow-up regardless of treatment change or discontinuation.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 67 | 78
percentage change | -1.41 [-3.78 to 0.00] | -2.91 [-4.84 to -1.06]

3. Secondary Outcome: Number of Participants With Primary Adverse Events
Description: Primary adverse events include all SAEs defined according to ICH guidelines and targeted protocol events, which include all diagnoses of hypercalcemia, hypophoatemia, and nephrolithiasis as well as signs and symptoms grade 2 or higher that may be associated with hypercalcemia and all laboratory toxicities grade 2 or higher defined by the 2004 DAIDS grading table
Time Frame: From first study treatment to week 48
Population: All enrolled subjects including subjects excluded from efficacy analysis due to eligibility violation.
Measure: Number; unit: participants
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 81 | 86
participants | 50 | 53

4. Secondary Outcome: The Change in Total 25-OH Vitamin D Level From Baseline to Weeks 24 and 48
Description: Changes in total 25-OH vitamin D from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
  Total 25-OH vitamin D is the sum of vitamin 25-OH D2 and D3 levels. All 25-OH vitamin D2 or D3 values below the lower limit of 1.25 ng/mL were imputed to 0 ng/mL
Time Frame: Weeks 0, 24, and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=71 and 74 for changes at week 24, n=65 and 68 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 71 | 74
ng/mL
  change from baseline to week 24 | 27.5 [15.0 to 38.0] | -0.8 [-5.9 to 4.9]
  change from baseline to week 48 | 24.2 [14.3 to 35.8] | 0.6 [-6.1 to 4.3]

5. Secondary Outcome: The Changes From Baseline in IL-6 to Weeks 24 and 48
Description: Interleukin 6 (IL-6) changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=66 and 68 for changes at week 24, n=58 and 62 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 66 | 68
log10 pg/mL
  change from baseline to week 24 | -0.05 [-0.23 to 0.11] | -0.04 [-0.23 to 0.14]
  change from baseline to week 48 | -0.07 [-0.24 to 0.12] | -0.03 [-0.23 to 0.10]

6. Secondary Outcome: The Changes From Baseline in sCD14 to Weeks 24 and 48
Description: Soluble cluster of differentiation 14 (sCD14) changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=68 and 68 for changes at week 24, n=62 and 63 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 68 | 68
log10 ng/mL
  change from baseline to week 24 | 0.02 [-0.08 to 0.15] | 0.00 [-0.07 to 0.14]
  change from baseline to week 48 | 0.07 [-0.05 to 0.16] | 0.02 [-0.06 to 0.14]

7. Secondary Outcome: The Changes From Baseline in P1NP to Weeks 24 and 48
Description: P1NP (marker of bone formation) changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=72 and 77 for changes at week 24, n=66 and 72 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 72 | 77
ng/mL
  change from baseline to week 24 | 11 [2 to 26] | 21 [12 to 38]
  change from baseline to week 48 | 15 [0 to 29] | 18 [7 to 39]

8. Secondary Outcome: The Changes From Baseline in CTX to Weeks 24 and 48
Description: CTX (marker of bone resorption) changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 72 | 77
ng/mL
  change from baseline to week 24 | 0.11 [-0.01 to 0.27] | 0.22 [0.11 to 0.35]
  change from baseline to week 48 | 0.10 [-0.04 to 0.25] | 0.14 [0.05 to 0.32]

9. Secondary Outcome: The Changes From Baseline in HOMA-IR to Weeks 24 and 48
Description: Homeostatic model assessment insulin resistance (HOMA-IR) changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=69 and 73 for changes at week 24, n=64 and 69 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: HOMA-IR
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 69 | 73
HOMA-IR
  change from baseline to week 24 | 0.17 [-0.21 to 0.91] | 0.39 [-0.11 to 1.15]
  change from baseline to week 48 | 0.13 [-0.26 to 1.11] | 0.26 [-0.44 to 0.79]

10. Secondary Outcome: The Changes From Baseline in Fasting Total Cholesterol to Weeks 24 and 48
Description: Fasting total cholesterol changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=74 and 80 for changes at week 24, n=68 and 73 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 74 | 80
mg/dL
  change from baseline to week 24 | 11 [-4 to 29] | 18 [1 to 31]
  change from baseline to week 48 | 13 [-6 to 28] | 14 [-1 to 37]

11. Secondary Outcome: The Changes From Baseline in Fasting LDL to Weeks 24 and 48
Description: Fasting LDL cholesterol changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=70 and 72 for changes at week 24, n=65 and 67 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 70 | 72
mg/dL
  change from baseline to week 24 | 0 [-10 to 17] | 8 [-11 to 20]
  change from baseline to week 48 | 2 [-9 to 14] | 4 [-14 to 27]

12. Secondary Outcome: The Changes From Baseline in Urinary Phosphate Excretion to Weeks 24 and 48
Description: Fractional excretion of phosphate changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
  Fractional Excretion of Phosphate (in %) is defined as:
  [Urine Phosphate x Serum Creatinine] / [Urine Creatinine x Serum Phosphate] x 100%
Time Frame: Weeks 0, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=58 and 70 for changes at week 24, n=59 and 69 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 58 | 70
percent
  change from baseline to week 24 | 0.7 [-2.4 to 3.1] | 0.2 [-1.8 to 3.8]
  change from baseline to week 48 | 0 [-1.8 to 3.7] | 0.9 [-1.9 to 4.0]

13. Secondary Outcome: The Changes From Baseline in CD4 to Weeks 4, 12, 24 and 48
Description: Total CD4 count changes from baseline to weeks 4, 12, 24 and 48 [week 4/12/24/48 - baseline].
Time Frame: Weeks 0, 4, 12, 24 and 48
Population: Included all available data regardless of treatment change/discontinuation, but was limited to eligible subjects who had both baseline and follow-up data.
  n=78 and 86 for changes at week 4, n=77 and 85 for changes at week 4, n=76 and 84 for changes at week 24, n=69 and 80 for changes at week 48.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 78 | 86
cells/mm^3
  change from baseline to week 4 | 74 [2 to 146] | 60 [15 to 102]
  change from baseline to week 12 | 103 [41 to 170] | 106 [60 to 216]
  change from baseline to week 24 | 138 [46 to 195] | 136 [66 to 219]
  change from baseline to week 48 | 192 [113 to 305] | 201 [108 to 292]

14. Secondary Outcome: The Changes From Baseline in iPTH to Weeks 24 and 48
Description: iPTH (Parathyroid Hormone, intact) changes from baseline to weeks 24 and 48 ( [week 24-baseline] and [week 48 - baseline], respectively).
Time Frame: Weeks 0, 24 and 48
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Number analyzed (Participants) | 72 | 77
pg/mL
  change from baseline to week 24 | 0.4 [-3.8 to 5.7] | 4.2 [-0.8 to 9.3]
  change from baseline to week 48 | 1.1 [-4.0 to 6.1] | 5.2 [-0.7 to 12.6]

ADVERSE EVENTS:
Time Frame: From first study treatment to week 48
Description: Adverse events from patients' first study treatment date to off study date.
  medDRA version 16.1
Arm/Group | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF
Serious Adverse Events (participants affected / at risk) | 8/81 | 7/86
Other Adverse Events (participants affected / at risk) | 60/81 | 70/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF (N=81) | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF (N=86)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Vitamin D3 and Calcium Carbonate Plus EFV/FTC/TDF (N=81) | Arm B: Vitamin D3 Placebo and Calcium Placebo Plus EFV/FTC/TDF (N=86)
Nausea (Gastrointestinal disorders) | 5 | 3
Alanine aminotransferase abnormal (Investigations) | 5 | 2
Alanine aminotransferase increased (Investigations) | 3 | 9
Aspartate aminotransferase abnormal (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 9
Blood albumin decreased (Investigations) | 5 | 6
Blood calcium decreased (Investigations) | 4 | 5
Blood cholesterol increased (Investigations) | 24 | 26
Blood glucose decreased (Investigations) | 9 | 19
Blood glucose increased (Investigations) | 15 | 16
Blood phosphorus decreased (Investigations) | 22 | 23
Blood sodium decreased (Investigations) | 4 | 8
Low density lipoprotein increased (Investigations) | 15 | 22
Neutrophil count decreased (Investigations) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No